CLINICAL TRIAL: NCT03785548
Title: Utilization of the Mirror During Pelvic Exams: Does it Reduce Patient Vulnerability and Discomfort?
Brief Title: Utilization of the Mirror During Pelvic Exams
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 18-107
Record Dates: First submitted 2018-12-19; First posted 2018-12-24 (Actual); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-07

CONDITIONS: Pelvic Exam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mirror group: This group of patients agree to have the mirror pelvic exam, and they will undergo routine pelvic examination by a physician with the usage of a mirror in the room.
  Interventions: Other: Usage of a mirror
- No mirror group: This group of patients decline a mirror, and they will undergo the standard pelvic examination.

INTERVENTIONS:
Other: Usage of a mirror — using a mirror during the pelvic examination
  Groups: Mirror group

SUMMARY:
This is a prospective cohort study to determine if using a birthing mirror during the patient's pelvic examination decreases patients's degree of vulnerability and discomfort.

DETAILED DESCRIPTION:
In Obstetrics and Gynecology and its gynecologic subspecialties, the pelvic examination is routine practice for screening and diagnostic purposes. Nevertheless, due to their intimate nature, pelvic examinations may result in loss of control, embarrassment, discomfort and anxiety.

The mirror pelvic exam has been a proposed technique to decrease patient anxiety and improve comfort during an already uncomfortable examination. However, little research has focused on this modality to date.

The purpose of this study is to investigate whether the mirror pelvic exam decreases the level of vulnerability and discomfort experienced during the pelvic examination.

ELIGIBILITY:
Inclusion Criteria:

* New patients undergoing a pelvic exam performed by a physician at Cincinnati Urogynecology Associates, TriHealth

Exclusion Criteria:

* Existing patients
* Unwillingness to participate in the study
* Physical or mental impairment that would affect the subject's ability to visualize the mirror during examination or to complete questionnaires
* Inability to understand English

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All women 18 years of age to 80, who undergo pelvic exam by a physician at Cincinnati Urogynecology Associates, TriHealth will be approached for recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tam T, Crisp CC, Hill AM, Aldrich E, Ghodsi V, Yook E, Yeung J, Pauls RN. Utilization of a Mirror During Pelvic Examinations: Does it Improve the Patient's Experience? Female Pelvic Med Reconstr Surg. 2021 Mar 1;27(3):208-213. doi: 10.1097/SPV.0000000000000975. PMID 33620906

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mirror Group | No Mirror Group
Started | 73 | 74
Completed | 71 | 74
Not Completed | 2 | 0
Not completed — age > 80 | 1 | 0
Not completed — no Postop queries | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirror Group | No Mirror Group | Total
Number analyzed (Participants) | 71 | 74 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.99 (12.96) | 57.84 (13.86) | 55.95 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 74 | 145
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants checked all that apply
  Participants
    White | 62 | 66 | 128
    Black or African American | 10 | 5 | 15
    American Indian/Alaska Native | 2 | 0 | 2
    Asian | 1 | 0 | 1
    Prefer not to answer | 0 | 2 | 2
    missing | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 71 | 74 | 145

OUTCOME MEASURES:

1. Primary Outcome: Group Difference in Visual Analog Scale (VAS) on Level of Vulnerability
Description: VAS on vulnerability level will be measured after the pelvic exam, and group difference after controlling for baseline vulnerability, will be calculated. The VAS is a validated 100 millimeter scale with 'no vulnerability' represented as 0 mm and 'very vulnerable' equating to 100 mm.
Time Frame: 30 minutes after the pelvic exam
Population: There are 2 missing outcomes from Mirror group
Measure: Mean (Standard Error); unit: mm
Arm/Group | Mirror Group | No Mirror Group
Number analyzed (Participants) | 69 | 74
mm | 13.294 (1.854) | 16.145 (1.789)
Statistical Analysis 1: Comparison: Mirror Group vs No Mirror Group; Test type: Other; p = 0.270, ANCOVA; F(1, 140)=1.225; Mean Difference (Final Values) = 2.851, 95% CI 2-sided [-2.241 to 7.944], Standard Error of Mean 2.576

2. Primary Outcome: Group Difference in Visual Analog Scale (VAS) on Level of Pain/Discomfort
Description: VAS on discomfort level will be measured after the pelvic exam, and group difference after controlling for baseline discomfort level, will be calculated. The VAS is a validated 100 millimeter scale with 'no pain' represented as 0 mm and 'most pain' equating to 100 mm.
Time Frame: 30 minutes after the pelvic exam
Population: Each group has 1 missing outcome.
Measure: Mean (Standard Error); unit: mm
Arm/Group | Mirror Group | No Mirror Group
Number analyzed (Participants) | 70 | 73
mm | 19.683 (2.201) | 19.824 (2.154)
Statistical Analysis 1: Comparison: Mirror Group vs No Mirror Group; Test type: Other; p = 0.964, ANCOVA; F(1, 140)=0.002; Mean Difference (Final Values) = 0.141, 95% CI 2-sided [-5.983 to 6.266], Standard Error of Mean 3.098

ADVERSE EVENTS:
Time Frame: within 30 minutes after pelvic examination
Arm/Group | Mirror Group | No Mirror Group
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/74
Other Adverse Events (participants affected / at risk) | 0/71 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT03785548/Prot_SAP_000.pdf